CLINICAL TRIAL: NCT02196805
Title: A Bioequivalence Study Comparing a Single Oral Intake of an Imported PROBUCOL Tablet(Lorelco) With a Marketed PROBUCOL Tablet(Chang Tai) in Chinese Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Patiman Juma, Otsuka Beijing Research Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 009-09-801-01
Record Dates: First submitted 2009-08-25; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Chinese Healthy Volunteers
Keywords: bioequivalence; imported PROBUCOL table; Lorelco; marketed PROBUCOL tablet; Chang Tai
MeSH Terms: interventions — Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Group A: imported Probucol ( Lorelco)
- 2 (Experimental)
  Interventions: Drug: Group B: Marketed Probucol ( Chang Tai)

INTERVENTIONS:
Drug: Group A: imported Probucol ( Lorelco) — Group A: take imported Probucol( Lorelco) (250mg/tablet), Qd, P.O.
  Arms: 1
Drug: Group B: Marketed Probucol ( Chang Tai) — Group B: take Marketed Probucol(Chang Tai)(250mg/tablet), Qd, P.O.
  Arms: 2

SUMMARY:
This study compares the pharmacokinetics characteristics of a single oral intake of an imported PROBUCOL tablet(Lorelco)(1*250mg/tablet) with a marketed PROBUCOL tablet (Chang Tai)(1*250mg/tablet) in healthy male volunteers to demonstrate they are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Male, aged between 18 and 40 years (at time of informed consent), extremes included
* Non-smokers
* Normal weight as defined by a Quetelet body mass index range of 18.0 - 26.0 kg/m2, extremes included
* Subjects judged by the investigator or sub investigator to be healthy based on the physical examination, medical history, vital signs, electrocardiogram (ECG), and the results of clinical laboratory tests
* Provided signed informed consent prior to beginning protocol-specific procedures, indicating that they understood the purpose of this study
* Willing to adhere to the study procedures described in this protocol

Exclusion Criteria:

* History of respiratory system disease, cardiovascular disease, Renal and Urogenital Disease, Gastrointestinal disease, hematological disease, Neuropsychiatric disease, endocrine diseases, hepatic disease or any other disease or physical condition which could have interfered with the interpretation of the study results
* Known hypersensitivity history to any prescription drug or over-the-counter medication
* Use of the following medications or products during the periods specified below:

Any medication within 14 days prior to scheduled study drug administration; Alcohol and caffeine within 7 days prior to scheduled study drug administration; Grapefruit or grapefruit products within 14 days prior to scheduled study drug administration

* Participation in any other clinical trial within 12 weeks prior to scheduled study drug administration, or intention to participate any other clinical trial during the course of the study
* Significant loss or donation of blood or plasma (200 mL) within 30 days prior to the start of the study
* Body weight <50kg
* History of drug abuse within past 5 years or positive urine drug screen results
* Subjects who test positive in HIV,HCV antibody,HBS antigen
* Otherwise judged by the investigator to be inappropriate for inclusion in the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
BE parameters: AUC0-t | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration.
BE parameters: Cmax | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters: Cmax | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration.
Pharmacokinetic Parameters: Tmax | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration
Pharmacokinetic Parameters: AUC0-t | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration
Pharmacokinetic Parameters: AUC0-∞ | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration
Pharmacokinetic Parameters: t1/2 | blood sample will be collected at 4,8,12,16,24,36,48,72,96,144,216,288,360,456,552,648 hour of drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Pei Hu, Dr., Principal Investigator — Clinical Pharmacology Research Center Peking Union Medical College Hospital
Locations (1):
- Clinical Pharmacology Research Center Peking Union Medical College Hospital, Beijing, China